Growth Mindset Psychoeducation for Modifiable Risk Factors for CMD NCT03707522 05/31/2018

#### **Research Integrity**

218 Ross Hall / 331, Reno, Nevada 89557 775.327.2368 / 775.327.2369 fax www.unr.edu/research-integrity

# Part II Application - Social Behavioral/Education Research

| Not | te the following: | |
|---|---|---|
| | <ol> <li>A Part I Cover sheet is required for each project submitted in IRBNet; see <u>Locating the Cover Sheet</u></li> <li>See IRB policy for submission requirements for new projects for <u>Full Committee Review</u> or <u>Expedited Review</u>.</li> </ol> | |
| PI F | Responsibilities Responsibilities Responsibilities | |
| 1. | How will the PI ensure that all study personnel are informed about the research plan and their research-related duties? | <ul> <li>X Routine meetings</li> <li>X Regular communication (e.g., email, phone)</li> <li>Other research staff training, describe:</li> </ul> |
| Stu | dy Sites and Collaborating IRBS | |
| 2. | List/describe the study sites: | University of Nevada, Reno |
| 3. | Will this research be reviewed by other IRBs? | X No Yes (Consider <u>contacting our office</u> for assessment and coordination of single IRB review.) |
| <u>Sel</u> | ection of Research Participants | |
| 4. | How many participants (or records) will be enrolled? | 500 Number of participants/records |
| 5.<br>X<br>—<br>X<br>—<br>6. | What are the participant eligibility inclusion criteric Age, specify: 18-65 years old Gender, specify: Race/ethnicity, specify: Language, specify: English Another country or specific culture , specify: Veteran status, specify: What are the participant exclusion criteria? | <ul> <li>Adults with cognitive impairmentill</li> <li>Pl's students, patients, or employeesiv</li> <li>Economically/educationally disadvantaged personsv</li> <li>Socioeconomic factors, specify: <ul> <li>Additional, describe:</li> <li>N/A, no exclusion criteria</li> <li>Description: Under the age of 18, not fluent in</li> </ul> </li> </ul> |
| 7. | Justify exclusions based on age, gender, or race: Will the research involve researchers' clients, | English. N/A, no such exclusions Justification: Minors will not be included as freshmen at orientation will likely not have a guardian present to provide informed consent. Non-English speakers will not be included in the study as translations of the material and measures are not available. Individuals over the age of 65 will not be included because risk factors for older adults may differ in important ways that would affect the content of the intervention material (e.g., Beekman, 1995) X No |
| ο. | students, or employees; or persons who are educationally or economically disadvantaged (see | Yes, specify and describe additional precautions to ensure participants are fully informed and |

| Red | Recruitment Methods and Materials | | | |
|---|---|---|---|---|
| | Check here if there are no proce | esses/mechanisms | to recruit participants; skip to | next section. |
| 9. | Who will recruit prospective particles and bow take place: | | Recruitment exclusively the PI X Co-investigators Study coordinator Research assistants Third party, specify and de relationship to the study pother, specify: N/A, recruitment exclusive Description of recruitment pro- | escribe the party's population: ely through SONA pocess: Participants will |
| | | | be recruited from freshmen or will be provided with a recruit provided by freshmen orienta. Research staff will also be pretable with flyers to provide infestudy. | ment flyer in the binder<br>tion programming staff.<br>sent at orientation at a |
| 11. | What <u>recruitment materials</u> will be used? <sup>vi</sup> | X Flyers/advert Emails/letters Scripts Slide or comp | Social m List servouter presentation X Other, socientation | nedia, specify: |
| Ass | sessing Participants for Eligibility Check here if participants will N | | r eligibility: <b>skip</b> to next section | |
| 12. | How will researchers confirm pa<br>eligibility for the research? | | Participants will complete a sequestions to ensure that tages of 18-65, fluent in Enfreshmen. | et of demographic<br>hey are between the |
| 13. | How will researchers inform par the process to assess eligibility? | ticipants about | Eligibility information will be in consent and study flyer. | ncluded in the informed |
| 14. | What will happen to screening/e individuals who are not eligible | | Screening/eligibility data for in eligible to participate will be drecruitment is complete. | |
| Recruitment Incentives/Payments | | | | |
| X Check here if there are no recruitment incentives/payments; skip to next section. | | | | |
| 15. | What types of recruitment incer will researchers give participant | | X Credit through SONA: .5 Soup up Course credit; equivalent, opportunities must be ava Money or gift cards; specify Raffle or drawing; specify winning: Other: specify and value: | alternative<br>iilable<br>fy amount: |

| 16. | When and how will researchers distribute | X SONA credit awarded via standard procedures | |
|---|---|---|---|
| | incentives/payments? | Description: | |
| 17. | For all incentives/payments, explain why the | X SONA credit, standard amounts | |
| | amount or value is reasonable for the research: | Explanation: | |
| 18. | Will participants be required to provide <i>Protected</i> | X No | |
| | Personally Identifiable Information (PPII) | Yes, specify the PPII required for payment, to | |
| | including social security numbers, to receive | whom it will be provided, and how it will be | |
| | incentives/payments? <sup>ix</sup> | protected during this process: | |
| Info | ormed Consent Methods/Procedures | | |
| | Check here if you do not plan to obtain informed of | onsent from participants); skip to the next section. x | |
| 19. | Describe the process for obtaining legally | N/A, research only involves children <sup>xi</sup> | |
| | effective informed consent from <i>each</i> participant | N/A, research only involves adults with impaired | |
| | (i.e., describe when, where, and how each recruit | consent capacity and surrogate consent <sup>xii</sup> | |
| | will be told about the research and agree to | Description of informed consent process: All | |
| | her/his participation). | freshmen completing orientation receive a binder as | ; |
| | | part of orientation programming. This binder | |
| | | contains information and resources for freshmen | |
| | | students. This binder will contain a study flyer that | |
| | | contains a brief description of the study. Research | |
| | | staff will also be present at an information table at | |
| | | orientation. If participants are interested in learning | |
| | | more, they can choose to access the Qualtrics site | |
| | | through a survey link provided in the flyer. If they | |
| | | choose to access the Qualtrics survey link, they will | |
| | | be able to read the informed consent prior to | |
| | | agreeing to participate in the study. | |
| 20. | Specify which researchers will obtain informed | X Via online or electronic information sheet | |
| | consent from participants: | — Pl | |
| | | <ul><li>Co-investigators</li><li>Study coordinator</li></ul> | |
| | | Research assistants | |
| | | Other, specify: | |
| 21. | How will researchers ensure consent is obtained | Check all that apply: | |
| | in a language understandable to participants? | X Consent materials reflect the expected literacy of | of |
| | | the sample population | |
| | | X Participants speak English | |
| | | Researcher fluent in participants' language will | |
| | | interpret | |
| | | Person in community will interpret | |
| | | Professional interpreter will be present | |
| | | Consent materials translated in participants' | |
| | | language or short-form consent process used | |
| | | Other, specify: | |
| 22. | How will researchers ensure individuals have | Participants will have as much time as they would lik | æ |
| | sufficient opportunity to consider participation? | to review consent materials. | |

No incentives will be offered for the first portion of 23. How will researchers protect participants from undue influence/coercion during the consent the study taking place during orientation. process? Participation in the follow-up assessment will be compensated using SONA credits. Participants may decline to participate in the study and participate in another research study in order to obtain credits. 24. How will researchers assess each person's As recommended by the IRB comprehension of the research? Other, specify: **Documentation of Consent** 25. Will participants sign an IRB-approved consent N/A, minimal risk research that is NOT conducted/supported by a federal agency form, as required at 45CFR46.117? (including the VA); and does NOT involve incomplete disclosure or deception, or prisoners No, requesting IRB approval to waive requirement for documentation of consentxiii Yes, via short form consent documentation (for non-English-speaking participants) **Research Costs** 26. Will participation result in out of pocket expenses X No (including costs for cell phones used in research), Yes, complete the following: co-pays, 3<sup>rd</sup> party payer costs, or research-related What costs will participants or 3<sup>rd</sup> party cover? injury costs?xiv What costs will the researchers cover? What costs will the VA cover? What costs will the sponsor cover? Study Design/Research Methods Describe in non-technical terms. 27. What is the background information that The present study intends to determine the effect of supports this research? (Summarize previous psychoeducation on engagement with modifiable risk work and provide references.) factors for depression and anxiety. While psychoeducation, and etiological beliefs about depression in particular, have been conceptualized as an important part of mental health literacy (MHL), little evidence exists to suggest what the content of psychoeducation should entail in order to improve the stated goals of MHL of recognition, management and prevention of common mental health problems such as anxiety and depression (Kelly, Jorm & Wright, 2007). As such, factors that increase both engagement with modifiable risk factors are key to the prevention of common mental disorders such as anxiety and depression. Risk factors are variables that if present increase likelihood of developing disorder. Modifiable

risk factors are those variables that could be reasonably altered by the individual without outside intervention). For depression and anxiety, these include health behaviors such as drug and alcohol use, weight management, coping strategies, sleep, positive activities, physical activities and social support (Cairns et al., 2014; Zimmermann, Chong, Vechiu & Papa, 2017).

Prevention is especially warranted for college students, because they are at a developmentally unique time of life before which 80% of individuals have not yet developed anxiety or depression. With respect to onset of depression, 20% of those with depression experience their first symptoms at age 19, meet criteria by age 25, 50% meet criteria by age 25, meet criteria by 38. Thus, college freshmen are at a key stage before which most individuals will have developed a disorder (Munoz, Mrazek & Haggerty, 1996).

Growth mindset may be an important aspect of preventative psychoeducation. Dweck and colleagues' (1995) cognitive model of motivation has generated a significant body of work demonstrating that individuals have "implicit theories," related to the malleability of a trait, and that individuals set goals and behave with respect to that aspect. Thus, learned concepts about the mutability of a trait have consequences for future behavior, and persistence on challenging tasks in particular. Mueller and Dweck (1998) show that children who receive praise for intelligence are more likely to exhibit behaviors of entity theorists by choosing easier tasks and spending less time on challenging problems, whereas children praised for efforts are more likely to resemble incremental theorists by choosing mastery goals and working through difficult problems. Beliefs about the malleability of self-attributes are learned and apply to specific traits. For example, an individual may have learned that intelligence is fixed but that a personality trait such as hostility is flexible (Yeager & Dweck, 2012; Scott & Ghinea, 2014). With respect to mental health, research on malleability beliefs has been limited, but it does appear that engendering a "growth mindset," is effective for the reduction of mental health problems (Schleider & Weisz, 2016).

Accordingly, beliefs about the malleability of emotions have been shown to predict depression outcomes in a sample of college students, with students endorsing beliefs in emotion malleability experiencing fewer symptoms of depression (Tamir et al., 2007). One possible mechanism through which this protective may occur is through the engagement with modifiable risk factors. Thus, research is needed to further demonstrate the effectiveness of growth mindset for the prevention of depression and anxiety, and to determine through what mechanism this intervention may be effective. 28. State the study purpose, research hypothesis, or The present study aims to determine the effect of research questions: presenting psychoeducation emphasizing "growthmindset," and information on modifiable risk factors on engagement with modifiable risk factors. We hypothesize that psychoeducation emphasizing that mental health is malleable will increase the participant's engagement with risk factors outlined in the intervention. Participants will randomly be assigned to complete one of four conditions: (1) Growth mindset + Modifiable risk factor information (2) Control + Modifiable risk factor information (3) Control + Growth mindset (4) Control + Control This design will allow assessment of the incremental effects of growth mindset and modifiable risk factor information as well as interactions between these conditions. We hypothesize that condition 1 will be associated with the greatest increase in engagement with modifiable risk factors for depression and anxiety followed by conditions 2-3 which will be associated with greater increases in engagement with modifiable risk factors than the control group (condition 4). 29. When appropriate (e.g., community-based N/A, not necessary/appropriate to involve participatory research, international research), community members how will you involve community members as Describe: advisors in the design/implementation of the research, and dissemination of results?

| 30. | Check all research methods/procedures that apply | to this research: |
|---|---|---|
| | Psychological or behavioral | Needs assessment research |
| | interventions/treatments | Program evaluation research |
| | Educational activities/interventions | Observational research |
| | Experimental-control group assignment | X Surveys, interviews, focus groups |
| | Cross-over design | Collection of data from records |
| | Computerized simulations | Retrospective |
| | Equipment/devices <sup>xv</sup> , specify: | Prospective |
| | Ethnographic research | Other, specify: |
| 31 | Which of these methods/procedures are | The article containing psychoeducation related to the |
| 31. | experimental (i.e., conducted to evaluate | mental health will be experimentally |
| | | • |
| | safety/efficacy or other outcomes)xvi? | manipulated. Participants will be randomly |
| | | assigned to one of four conditions. |
| | | (1) Crowth mindest & Madifiable rick factor |
| | | (1) Growth mindset + Modifiable risk factor |
| | | information |
| | | (2) Control + Modifiable risk factor information |
| | | (3) Control + Growth mindset |
| | | (4) Control |
| 22 | Which of these methods/procedures are | Neither procedure is considered usual care. |
| 32. | considered standard-of-care? | Neither procedure is considered usual care. |
| 22 | Who will provide the standard treatment or care | X N/A, research does not include usual |
| 33. | referenced above? | care/standard treatment |
| | referenced aboves | - |
| | | Study team |
| | | Participant's own health care provider |
| 2.4 | NA/less in grown agains are and a consequence and heavy will | Other, specify |
| 34. | Why is group assignment necessary, and how will | N/A, research does not involve group assignment |
| | participants be assigned to | Justification/description: Group assignment is |
| | treatment/experimental or control groups? | necessary to determine the differential effect of |
| | | each article on task engagement and persistence. |
| | | Participants will be randomly assigned to a |
| | | condition using Qualtrics survey software. |
| 35. | What will participants experience or be asked to | In all conditions, participants will be asked to read an |
| | do when assigned to the treatment / | article about mental health and complete a battery of |
| | experimental group <i>or</i> to the control group? | questionnaires at Time 1. In both conditions, |
| | | participants will complete a battery of questionnaires |
| | | at Time 2 and Time 3. |
| 36. | Note the expected number/length of | 3 Expected number of contacts/meetings |
| | contacts/meetings, and time commitment for | Minutes/hours for each contact/meeting |
| | participation (include similar information in | 30 minutes at Time 1 |
| | consent materials): | 15 minutes at Time 2 |
| | | 15 minutes at Time 3 |
| | | Duration of participation (in |
| | | weeks/months) for intervention |
| | | 30 minutes for intervention |

Duration of participation (in weeks/months) for long-term follow-up Follow up at Time 2 (one week following Time 1) Follow up at Time 3 (during Fall semester, 3-4 months following Time 1) **Data Collection and Analysis** 37. List the information/specimens that researchers Information collected will be data from the battery of will obtain for this research xvii: questionnaires at Time 1, Time 2 and Time 3. At Time 1, participants will be provided with a participant ID number. Participants will provide their e-mail address at this time. Participant ID will be stored in a file with the participant's e-mail address for follow-up contact purposes. 38. How will research data be obtained?xviii Research data will be obtained through Qualtrics survey software. 39. Identify each research instrument (e.g., diary, <u>Demographic questions</u>. Participants will be asked questionnaire, data collection log) and describe their gender, age, marital status, race/ethnicity, level of education and treatment seeking history and how its use relates to the study purposexix: intent. Patient Health Questionnaire. Severity of depression will be measured via the Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer & Williams, 2001), a 9-item questionnaire associated containing one item for each symptom of MDD as specified by the DSM. The PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for MDD. This measure has demonstrated good internal reliability ( $\alpha$ =.86). GAD-7. Anxiety severity will be measured using the Generalized Anxiety Disorder 7-item scale (GAD-7; Spitzer, Kroenke, Williams & Lowe, 2006) is a common, brief measure of anxiety symptom severity  $(\alpha = .92;).$ ARM-CMD. Mental health literacy will be assessed using the Awareness of Risks and Management of Common Mental disorders (ARM-CMD) measure developed to assess knowledge and attitudes related to the effective recognition, management and prevention of mental disorders (Zimmermann et al., in preparation). SF-36- Physical and Mental Health Short Forms. This measure includes sleep, social activity and health subscales. Sub-scales vary in response formats with

items rated from either 1-6 or 1-5 (Tarlov et al., 1989). Healthy diet questionnaire. Healthy diet will be assessed using a 10-item yes/no scale total of 10 points for health eating behaviors. Higher scores indicates that the participant tries to eat more fiber, more fruit, more vegetables, more fish, less meat, less sweets and pastries, tries to avoid the intake of fat, the consumption of butter, removes fat from meat does not add sugar to drinks (Zazpe et al., 2011). Substance Use Measure. Alcohol and substance use will be assessed using a 3-item substance use measure including frequency of alcohol use, cigarette use and drug use (Lee et al., 2015) The internal reliability estimate is  $(\alpha)$  .74. Brief COPE. Coping strategies will be assessed using the Brief COPE, a 28-item scale assessing various dimensions of healthy and unhealthy coping (B-COPE; Carver, 1997). Ryff Purpose in life scale. Purpose in life will be assessed using a 9-item scale (Ryff & Keyes, 1989). Mental health immutability beliefs measure. Immutability beliefs will be assessed after the manipulation is complete using a 4-item Likert scale from "strongly disagree," to "strongly agree." Items will be modified from the depression immutability beliefs questionnaire (Schroder et al., 2016) to refer to general mental health (e.g., "Your mental health is something about you that you cannot change very much.") SPSS will be utilized to conduct a 4 factor between 40. How will researchers analyze the data?<sup>™</sup> subjects ANOVA, to determine differences between groups in engagement with modifiable risk factors as well as to probe interactions between the effect of receiving the growth mindset education and information about modifiable risk factors. 41. Will this research include records of participants' No voices or images?xxi Yes, audio; describe and justify: Yes, video; describe and justify: Yes, photographs; describe and justify:

| Res | Research Risks | |
|---|---|---|
| 42. | Describe how risks will be minimized through use | X N/A, minimal risk research |
| | of sound research design: | Description: |
| 43. | What precautions will researchers use to avoid | Check all that apply: |
| | unnecessarily exposing participants to risk? | X N/A, minimal risk research |
| | | Using recognized standard practices |
| | | Ensuring researcher expertise/credentialing |
| | | Researcher training |
| | | Minimizing time required for procedures |
| | | Using procedures that are already being |
| | | performed (e.g., for education or treatment) |
| | | Monitoring participants for adverse reactions |
| | | Monitoring data for safety |
| | | Other, specify: |
| 44. | List the discomforts and physical harms that | No physical discomfort or harm is expected to |
| | might result from participation in this research; | result from participation in this study. |
| | assess the probability, severity, and duration of | |
| | each discomfort/harm: | |
| 45. | List the social, legal, financial, emotional, or | It is possible that emotional discomfort may |
| | familial harms might result from participation in | result from reading about mental health. It is |
| | this research; assess the probability, severity, and | unlikely that this emotional discomfort will |
| | duration of each of these harms: | persist after the completion of the study. |
| 46. | Identify secondary and incidental findings (see | X N/A, secondary/incidental findings not expected |
| | Policy Manual Definitions) that are reasonably | |
| | expected to result from this research. | |
| | Explain the plans for whether the findings to participants or others will be disclosed: | |
| 17 | How will participants be referred to | N/A, need for referrals not anticipated |
| 47. | psychological, or other services that may be | Explanation: All participants will be provided with a |
| | required as a consequence of participation in the | list of contact information for on-campus |
| | research? | psychological services including the Counseling |
| | | Services Center, Psychological Services Center and |
| | | Downing Clinic (see attached). |
| Saf | ety Monitoring for Greater than Minimal Risk Rese | |
| X | | ety monitoring is not required; skip to next section. |
| 48. | Describe the plan to monitor data for safety. | |
| | Include: | |
| | Who will monitor the data for safety | |
| | concerns? | |
| | <ul><li>What data will be reviewed?</li></ul> | |
| | <ul> <li>How often will the monitoring occur?</li> </ul> | |
| | • How often will cumulative data be reviewed? | |
| 49. | Are there specific findings that would trigger an | No |
| | immediate suspension of the research? | Yes, specify: |

| Res | search Benefits | | |
|---|---|---|---|
| 50. | Are individual participants expected to benefit from being in this research? | X | No: It is possible that the individual may benefit from learning more about mental health, but these benefits are not certain. Yes, specify: |
| 51. | What is the potential value of the knowledge to be gained from this research? | vali<br>psy<br>lite<br>me<br>wit | e knowledge gained from this research would be uable in determining what should constitute core rchoeducation components of mental health racy interventions in ways that serve to promote ntal health through the increased engagement h modifiable risk factors to prevent anxiety and pression. |
| <u>Pro</u> | tecting Participant Privacy | | |
| 52. | Will Protected Personally Identifiable Information (PPII) be collected for this research (see Policy Manual Definitions)? | х<br>— | No<br>Yes, specify what PPII will be collected and why it<br>is necessary to collect it: |
| 53. | How will researchers protect the privacy of prospective participants during initial contact, and interventions or interactions? | pas | a will be de-identified stored on a secure ssword protected computers that will only be illable to the PI and study personnel. |
| 54. | What protections will be in place for investigators to access records generally considered private (e.g., education or personnel records)? | x<br> | N/A, records generally considered private will not<br>be accessed for the research<br>Compliance with FERPA (for education records)<br>Other, describe: |
| 55. | Do any state laws for mandatory reporting apply to this research? (See IRB policy for applicable Nevada State Laws.) | X<br>— | No<br>Yes, specify and include in consent document: |
| 56. | For researching involving the collection of identifiable information that may have legal ramifications (e.g. illegal drug use, criminal activity), will a <i>Certificate of Confidentiality</i> be obtained (see <a href="IRB CoC policy">IRB CoC policy</a> )? | <br>X<br> | N/A, no such information will be collected N/A, identifiers not collected or not maintained No, explain why not: Yes, upon receipt of the COC, create a new package, and Add the certificate. |
| Ma | intaining Data Confidentiality | | |
| 57. | Identify the formats in which research records will be maintained by the PI: | <br> | Paper Electronic Recorded media (e.g., audio/video, digital photos) Other, specify: |
| 58. | 58. Where will research records be maintained by the PI?xxii (Check all that apply.) | | |
| X<br> | Password-protected file on University/Affiliate server (e.g., UNRNAS) or secure VA network server In the UNR Med-hosted environment On an external cloud-based solution; Add | <br> | In a locked file cabinet in the PI's office or lab In a locked or password-protected office or lab at the University, Affiliate site, or VASNHCS Off-site in a secure facility with password- protected access, <b>Add</b> Business Associate |
| | Business Associate Agreement or ORD approval for VA research | _ | Agreement VA research only, off-site in another VA facility, specify: |

| | On a password-protected stand-alone | | VA research only, off-site in a secure non-VA |
|---|---|---|---|
| | desktop/laptop computer (must be encrypted) | | facility with password-protected access, Add |
| | On a password-protected Electronic Portable | | documentation of ORD approval |
| | Device (must be encrypted) | | Other location, specify: |
| 59. | Who will have access to research records? | Che | eck all that apply: |
| | NOTE: It is understood the US DHHS, and UNR RI | Х | Principal Investigator |
| | and IRB will have access. | Х | Co-Investigators |
| | | | Research assistants |
| | | | Collaborating researchers, institutions or |
| | | | organizations, specify: |
| | | | Study sponsor |
| | | | VASNHCS or Affiliate Site Research Office |
| | | | Other federal agencies, specify: |
| | | | Other, specify: |
| 60. | How will researchers protect against | | N/A, data will be collected without identifiers |
| | unauthorized disclosure of identifiable | | Data will immediately be stripped of personal |
| | information about participants? | | identifiers; no master code list |
| | | Х | Data will be coded; master code list will be stored |
| | | | securely and separately |
| | | | Other, specify: |
| 61. | Will web-based applications be used to obtain, | | No |
| | record, or store data (e.g., online survey | Χ | Yes, identify the server/application xxiii Qualtrics |
| | administrator or sponsor-portal)? | | |
| 62. | Will software provided by a 3 <sup>rd</sup> party (e.g., | Х | No |
| | sponsor) be used to record or transmit data? | | Yes, identify the software and the source; |
| | | | summarize or <b>Add</b> data security policy: |
| 63. | Will mobile devices be used to collect or record | Х | No |
| | data for this project? | | Yes, with FIPS 140-2 encryption standard |
| | | | Yes, with other security measures, specify: |
| 64. | Will identifiable research records be transmitted | Χ | No |
| | or shipped to another location/institution? | | Yes, describe how confidentiality will be |
| | | | maintained during transmission/shipping: |
| 65. | How long will the PI store identifiable records? | | N/A, identifiers not collected or not kept |
| | | | N/A, data coded; master list will be destroyed |
| | | | before permanent storage |
| | | Χ | Until the study closes |
| | | | Years after study closure (note number): |
| | | | Indefinitely |
| | | | Other, specify: |
| 66. | What will happen to identifiable records after the | stor | age period ends? (Check all that apply.) |
| | N/A, identifiable data not collected or not stored | | Coded data will be placed in an existing |
| | N/A, research data and records will be stored | | repository; master code list will be destroyed |
| | indefinitely (per VHA Records Control Schedule | | Coded data will be placed in an existing |
| | 10-1 when applicable) | | repository; master code list will be maintained by |
| | Paper/electronic records will be destroyed. | | the repository |
| | Audiotapes/videotapes will be erased or | | Data along with PPII will be maintained by the PI |
| | destroyed | | for future research purposes |

| Х | The master code list will be destroyed; de-<br>identified data will be maintained by the<br>Investigator indefinitely | Other, describe: |
|---|---|---|
| Tra | insferring Research Data to a Bank or Repository fo | or Future Uses |
| X | Check here if this is data will not be transferred to | o a bank or repository; skip to next section. |
| 67. | Will <i>identifiable</i> research data be transferred to a data bank or repository for future use? NOTE: Information about future uses <i>must</i> be in consent documents. | <ul> <li>No</li> <li>Yes, name the bank/repository, justify the retention of identifiers, and describe future uses:</li> </ul> |
| 68. | Specify the oversight mechanisms for future uses of identifiable data transferred to a bank/repository: | <ul> <li>N/A, identifiable data will not be transferred to a bank/repository</li> <li>Existing repository has appropriate oversight mechanisms in accordance with VHA Handbook 1200.12.</li> <li>IRB of Record for the bank/repository is responsible for approval and oversight of research involving the records</li> <li>Other, specify:</li> </ul> |
| Ad | ditional Requirements for VA Research | |
| Χ | <b>Check here</b> if this is not VA research; <b>skip</b> to next s | ection. |
| 69. | Check the employment category that applies to the Principal Investigator: | <ul> <li>VA employee, specify VA percentage of time in 8<sup>ths</sup>:</li> <li>VA WOC (Without Compensation)</li> <li>VA-contracted personnel</li> <li>Other, specify:</li> </ul> |
| 70. | How is this research relevant to Veterans? | |
| 71. | If the research involves non-Veteran participants, describe VA's coverage of costs resulting from research-related injury: | N/A, all participants will be Veterans Description: |
| 72. | Will a non-VA entity (other than as disclosed above) have access to VA-Sensitive Information/Data (as defined in VA Handbook 6500, Appendix A)? | <ul> <li>No</li> <li>Yes, name the entities and check the type of agreement that will be in place, and Add a copy of the agreement: <ul> <li>Data Use Agreement</li> <li>Cooperative Research and Development Agreement (CRADA)</li> <li>Other, specify:</li> </ul> </li> </ul> |
| Inf | ormed Consent Documents/Materials | |
| | Check here if you request IRB approval to waive the | e requirement for informed consent and skip section. |
| 73. | What materials will be used to inform participants about the research?xxiv | <ul> <li>N/A, not obtaining consent</li> <li>Sponsor consent template, revised using Consent Checklist</li> <li>Consent form or information sheet based on a Consent Form Template from IRBNet</li> </ul> |

| | | | Simplified info script, sheet, email, letter based on a <i>Consent Information Script/Sheet Template</i> from IRBNet Other, specify: |
|---|---|---|---|
| 74. | Will participants in <i>greater than minimal risk</i> research be provided with the DHHS required basic and additional elements of informed consent (as specified at 45CFR46.116)? | X<br>— | N/A, minimal risk research N/A, under IRB-Flex for greater than minimal risk research, elements that do not apply to the research are excluded Yes Ves Ves Ves Ves |
| 75. | Will participants in <i>minimal risk research</i> that is conducted/supported by a federal agency, or that involves <u>incomplete disclosure/deception</u> or prisoners be provided with the DHHS required basic and additional elements of informed consent (as specified at <u>45CFR46.116</u> )? | x<br> | N/A, greater than minimal risk research (addressed above) N/A, minimal risk research that does NOT involve federal funding, incomplete disclosure or deception, or prisoners N/A, PI requesting IRB approval for <i>alteration</i> of DHHS requirements for informed consent xxvi Yes, using a <i>Consent Form Template</i> from IRBNet to create the consent document |

### Obtain the electronic signature of Principal Investigator to confirm the following PI assurances:

#### **University/Affiliate Principal Investigator Assurance**

My electronic signature certifies that I have read/prepared the project documents and agree to comply with the <u>PI responsibilities in the IRB Policy Manual</u> and applicable Affiliate policies.

Obtain the electronic signature of a Responsible Official (RO) or Affiliate Representative.

## **University/Affiliate Responsible Official Assurance**

My electronic signature certifies that I have read the project documents, and agree to comply with the <u>RO</u> <u>responsibilities in the IRB Policy Manual</u> and applicable Affiliate policies.

Add copies of collaborating IRB decisions, as Other

ii **Add** form *Research*: *International* 

Add form Population: Persons with Cognitive Impairment

See IRB policy for inherently influential recruitment situations

See IRB policy for inherently influential recruitment situations

vi Add copies of all recruitment materials, as Advertisements.

vii **NOTE**: Data must be retained for VA research.

viii **Disclose** in consent materials, gift value and odds of winning.

ix Disclose in consent materials, requirement for participant to provide PPII to receive payment.

<sup>\*</sup> Add form Consent Waivers.

xi Add form Population: Children to describe child assent and parental permission

xii Add form Population: Persons with Cognitive Impairment

xiii Add form Consent Waivers.

viv **Disclose** costs to participants or 3<sup>rd</sup>-party payer in consent materials.

<sup>&</sup>lt;sup>xv</sup> **For example**: Retinal scans, skin galvanometers,

wi NOTE: All research components that are experimental must be identified as such in consent materials.

include information that will be obtained from existing records, from activities/procedures performed solely for the research, or from activities/procedures performed as part of standard treatment/educational practice.

include descriptions for obtaining data from existing records, prospectively from study procedures, or prospectively from procedures performed for standard treatment/educational practices.

xix **Add** non-standard instruments as *Questionnaire/Survey* or *Data Collection*, as applicable.

For multi-site research specify if site-specific data will be analyzed separately. If data will be pooled, indicate if participant identifiers will be maintained and describe how findings will be shared among cooperating PIs.

<sup>&</sup>lt;sup>xxi</sup> **ONLY** for video or photographs, **Add** video/photo release form. (Release form not required for VA research.)

See <u>University IT Data Management</u> on the web for information about electronic data management/storage solutions. Additional requirements apply to storage of identifiable information outside of the University. Investigators planning to store Identifiable data on a cloud-based solution or off-campus, *must* contact the University Chief Information Security Officer in the University IT office for requirements.

xxiii Add copies of the site's privacy/data security policies.

xxiv **Add** all consent materials.

xxv Use either the *Consent Checklist* to revise sponsor consent templates or a *Consent Form Template* from IRBNet to create a consent document.

xxvi **Add** form *Consent Waivers*.